CLINICAL TRIAL: NCT03982745
Title: Efficacy of Bonfils Fiberoptic Stylet for Tracheal Intubation With Double Lumen Tube After Failure of Direct Laryngoscopy. A Prospective Study
Brief Title: Double Lumen Tube Positioning With Bonfils Fiberoptic Stylet: Prospective Observational Study in 30 Adult Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Director, Università Politecnica delle Marche
Other Study IDs: 2018-335
Record Dates: First submitted 2019-05-30; First posted 2019-06-11 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Difficult Intubation; Thoracic Surgery
Keywords: bonfils fiberoptic stylet; double lumen intubation; thoracic surgery; difficult intubation; difficult airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: bonfils — bonfils intubation

SUMMARY:
The aim of this prospective observational study is to evaluate the efficacy of Bonfils fiberoptic stylet to perform tracheal intubation with double lumen tube after failure of standard laryngoscopy in 30 adults patients scheduled for elective thoracic surgery, who require tracheal intubation with double lumen tube for One Lung Ventilation under general anesthesia in a teaching hospital operating theatre at Ospedali Riuniti Ancona (Italy).

DETAILED DESCRIPTION:
This is a prospective, observational study, approved by Marche's Regional Ethics Committee (CERM), Ancona, ITA on the 07 February 2019. The study is conformed to the Declaration of Helsinki and Good Clinical Practice guidelines, an informed written consent will be obtained at recruitment.

The aim of this study is to evaluate the efficacy of Bonfils fiberoptic stylet to perform tracheal intubation with double lumen tube (DLT) after failure of standard laryngoscopy in 30 adult patients (patients 18 years of age) scheduled for elective thoracic surgery, who require tracheal intubation with (DLT) for One Lung Ventilation (OLV) under general anesthesia. The study will be performed in a teaching hospital operating theatre at AOU Ospedali Riuniti Ancona (Italy).

Pre-operative evaluation will be done before surgery, demographic variables will be collected and the clinical screening tests to predict a difficult airway will be performed.

On the day of the intervention, patients will be subjected to standard monitoring of vital signs (NIBP, FC, SpO2 and ECG) and, after induction of general anesthesia and adequate pre-oxygenation (3-minutes with facial mask ventilation), a direct laryngoscopy with Macintosh blade will be performed to insert a DLT. The Cormack-Lehane grade view will be registered after optimization of the intubation attempt by improving the "sniffing position" and the external manipulation of the larynx (BURP maneuver). In case of declaration of intubation failure, it will be used Bonfils fiberscope for the DLT insertion.

A maximum duration of intubation attempt is not established, but a decrease in SpO2 below 90% will be considered as a criterion for abandoning the procedure and the patient will be re-oxygenated.

The maximum number of attempts allowed will be 2 for the Macintosh laryngoscope and 2 for the Bonfils fiberscope, after which, in case of failure with the both devices, the patient will be awakened.

In any case of difficulty in patient oxygenation and ventilation with facial mask, a second generation laryngeal mask will be used. The following parameters relating to the patients recruited in the study will be recorded: weight, height, BMI, Mallampati score, interincisor distance, chin-Thyroid distance, Cormack-Lehane view grade at direct laryngoscopy.

The primary end point of this study is to assess the success rate of DLT insertion with Bonfils fiberscope.

The duration of the procedure, the number of attempts and the occurrence of any complications will also be recorded

Data analysis will be performed using the Medcalc 7.3.0.1 statistical program (Medcalc software, Ostend, Belgium). Kolmogorov-Smirnov's test will be used to test the normality of distribution.

Data will be presented as mean ± dev. standard or median and 95% confidence interval.

The results will be averaged, and the data will be presented as mean SD for each variable with continuous data. Values of P less than 0.05 will be considered as statistically significant.

The differences between means will be studied by parametric tests (eg Student's t) if the data are normal distribution and non-parametric tests (eg Wilcoxon) if the distribution is not normal.

With regard to the efficacy of Bonfils fiberscope, literature have been reported a success rate higher than 80%. Therefore, assuming a success rate of around 90% (and accepting a standard deviation of 10%), we should study at least 30 patients for whom we expect to have a correct tracheal intubation on about 27 patients. A 5% SD would mean that intubation will be successful in at least 26 patients (85%), which we believe could be considered an excellent result.

ELIGIBILITY:
Inclusion Criteria:

* adults (age≥18 years)
* tracheal intubation with double lumen tube (DLT) for One Lung Ventilation (OLV) required for elective thoracic surgery under general anaesthesia

Exclusion Criteria:

* patients undergoing emergency thoracic surgery
* patients with predictive criteria of difficult ventilation scheduled for "awake endoscopic intubation"
* patients with anatomical features that contraindicate direct laryngoscopy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults (patients 18 years of age) scheduled for elective thoracic surgery, who require tracheal intubation with double lumen tube (DLT) for One Lung Ventilation (OLV) under general anesthesia in a teaching hospital operating theatre at Ospedali Riuniti Ancona.
  Pre-operative evaluation will be done before surgery, demographic variables will be collected and the clinical screening tests to predict a difficult airway will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
the efficacy of Bonfils fiberoptic stylet to perform tracheal intubation with double lumen tube after failure of standard laryngoscopy | up to 2 minutes from device insertion
  the success rate of the procedure defined by the correct position of the double-lumen tube in the bronchial lumen verified by a flexible fiberscope

SECONDARY OUTCOMES:
Time to intubation, | up to 2 minutes from device insertion
  Time in minutes measured from device insertion into the patient's mouth until the DLT will be positioned into the bronchial lumen.
Any complications occurred | up to 12 hours measured from the insertion of the device
  number of patients that axperienced desaturation, hemodynamic alterations, oral cavity-pharynx and larynx traumatism
Number of intubation attempts | up to 15 minutes. The maximum number of attempts allowed will be 2 for the Macintosh laryngoscope and 2 for the Bonfils fiberscope, after which, in case of failure with the both devices, the patient will be awakened.
  number of attempt to intubation. intubation will be considered complete when the DLT will be positioned correctly into the bronchial lumen.

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, PhD, MD, Study Director — Università Politecnica delle Marche
Locations (1):
- AOU Ospedali Riuniti Ancona - Università Politecnica delle Marche, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No